CLINICAL TRIAL: NCT03743493
Title: PCORnet Opioid Surveillance Demonstration Project
Brief Title: PCORnet Opioid Surveillance Study
Status: Completed | Type: Observational
Sponsor: Louisiana Public Health Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Patient-Centered Clinical Research Network (Other); Research Action for Health Network (REACHnet) (Other); The Patient-Oriented Scalable National Network for Effectiveness Research (Other); ADVANCE Clinical Data Research Network (Unknown); New York City Clinical Data Research Network (Other); PaTH: Towards a Learning Health System Clinical Data Research Network (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency); Harvard Pilgrim Health Care (Other)
Responsible Party: Sponsor
Other Study IDs: OpioidRCR
Record Dates: First submitted 2018-10-26; First posted 2018-11-16 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Opioid Use; Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Prevalence numerator: An opioid prescribed or dispensed in the query period (1/1/2010-12/31/2017)
- Prevalence denominator: Any diagnosis on record in the query period (1/1/2010-12/31/2017)
- Guideline A numerator: An opioid prescribed or dispensed in the query period (1/1/2010-12/31/2017) AND NO cancer diagnosis in the year prior to the index event
- Guideline A denominator: Any diagnosis on record in the query period (1/1/2010-12/31/2017) AND NO cancer diagnosis in the year prior to the index event
- Guideline B numerator: An opioid prescribed or dispensed in the query period (1/1/2010-12/31/2017) AND NO inpatient cancer diagnosis OR cancer procedure in the year prior to the index event
- Guideline B denominator: Any diagnosis on record in the query period (1/1/2010-12/31/2017) AND NO in-patient cancer diagnosis OR cancer procedure in the year prior to the index event

SUMMARY:
The overarching objective of this project is to demonstrate and assess the feasibility of using the Patient Centered Outcomes Research Network (PCORnet) Common Data Model for opioid surveillance to complement existing and support future initiatives. This project will characterize risk factors, processes, and outcomes related to opioid use, misuse, and abuse. It will quantify the utility of data stored in the PCORnet Common Data Model format stewarded by healthcare organizations participating in PCORnet.

DETAILED DESCRIPTION:
This is a two phase retrospective study. The goal of Phase I is to assess the utility of PCORnet Common Data Mode (CDM) data to study risk factors, processes, and outcomes related to opioid use, misuse, and abuse. Based on the results of the Phase I feasibility examination, Phase II will be conducted and will analyze the relationships between patient- and provider-level risk factors and policies, and opioid-related outcomes over time and within geographic regions.

The study will leverage the existing data PCORnet data infrastructure and resources to achieve its objectives and answer its research questions. Standardized analysis programs will be distributed to participating sites within the PCORnet Distributed Research Network. Sites will return aggregate, descriptive counts and summary statistics from regression analyses. When data are unavailable or analysis is determined infeasible, results will be reported as such.

The Aims of Phase I are:

1. Generate counts and proportion of patients with exposure (or potential exposure) to opioids though prescription or dispensing records within a health system.

   a. Compare results to CDC.
2. Characterize data elements in PCORnet data and assess suitability for opioid surveillance.

   1. Identify the relevant data elements
   2. Examine data completeness and validity
   3. Identify data limitations and gaps that limit surveillance

The Aims of Phase II are:

1. Examine whether and to what extent patient-level risk factors, provider processes, and policies are associated with declines in outcomes of interest.
2. Examine whether and to what extent prescribing guidelines, related policies, processes, and/or care procedures are associated opioid-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

• Patients with an opioid exposure (prescription or dispense) or diagnosis from an encounter on record between 1/1/10-12/31/17.

Exclusion Criteria:

• Patients without an opioid exposure (prescription or dispense) or diagnosis from an encounter on record between 1/1/10-12/31/17.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with electronic health record data from participating clinical data research networks (CDRN) of PCORnet.
Sampling Method: Non-Probability Sample
Enrollment: 15438284 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Opioid exposure (prescribing/dispensing) counts by Guideline A group | 1/1/2010-12/31/2017
  Counts used to derive rates
Opioid exposure (prescribing/dispensing) counts by Guideline B group | 1/1/2010-12/31/2017
  Counts used to derive rates
Opioid exposure (prescribing/dispensing) counts by Prevalance group | 1/1/2010-12/31/2017
  Counts used to derive rates
Opioid exposure (prescribing/dispensing) counts stratified by demographic characteristics | 1/1/2010-12/31/2017
  Age group, sex, race and ethnicity; Counts used to derive rates
Most common diagnoses among cohort groups stratified by demographic characteristics and geography | 1/1/2010-12/31/2017
  Frequencies of most common 1000 diagnosis codes stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Most common procedures among cohort groups stratified by demographic characteristics and geography | 1/1/2010-12/31/2017
  Frequencies of most common 1000 procedure codes stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Occurrence of mental health diagnoses among cohort groups stratified by demographic characteristics and geography | 1/1/2010-12/31/2017
  Frequencies of mental health diagnosis codes stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Occurrence of opioid overdose diagnoses among cohort groups stratified by demographic characteristics and geography | 1/1/2010-12/31/2017
  Frequencies of opioid overdose stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Occurrence of substance use disorder diagnoses among cohort groups stratified by demographic characteristics and geography | 1/1/2010-12/31/2017
  Frequencies of substance use disorder diagnoses stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Opioid exposure (prescribing/dispensing) counts by cohort groups and provider | 1/1/2010-12/31/2017
  Stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Most common diagnoses in patients with opioid-inclusive substance use disorder diagnoses | 1/1/2010-12/31/2017
  Frequencies of most common 1000 diagnosis codes overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Most common procedures among patients with opioid-inclusive substance use disorder diagnoses | 1/1/2010-12/31/2017
  Frequencies of most common 1000 procedure codes overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Occurrence of mental health diagnoses among patients with opioid-inclusive substance use disorder diagnoses | 1/1/2010-12/31/2017
  Frequencies of mental health diagnosis codes overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Occurrence of urine drug screening in patients with opioid exposure (prescribing/dispensing) | 1/1/2010-12/31/2017
  Frequencies of urine drug screening procedures or lab codes overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of HIV diagnoses in patients with opioid use disorder diagnosis | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of Hepatitis B diagnoses in patients with opioid use disorder diagnosis | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of Hepatitis C diagnoses in patients with opioid use disorder diagnosis | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of opioid and benzodiazepine co-prescribing/dispensing | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of Naloxone administration during an emergency department encounter among patients with an opioid overdose diagnosis | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of Naloxone exposure (prescribing/dispensing) among patients with opioid exposure (prescribing/dispensing) by encounter setting | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of Naloxone exposure (prescribing/dispensing) among patients with opioid-inclusive substance use disorder diagnosis by encounter setting | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of buprenorphine exposure (prescribing/dispensing) among patients with opioid-inclusive substance use disorder diagnosis by encounter setting | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of naltrexone exposure (prescribing/dispensing) among patients with opioid-inclusive substance use disorder diagnosis by encounter setting | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Frequency of methadone exposure (prescribing/dispensing) among patients with opioid-inclusive substance use disorder diagnosis by encounter setting | 1/1/2010-12/31/2017
  Counts overall and stratified by age group, sex, race, ethnicity, and facility 3-digit zip code
Adjusted risk of overdose in patients with opioid exposure (prescribing/dispensing) | 1/1/2010-12/31/2017
  Patient level regression controlling for year, age, sex, race, ethnicity
Adjusted risk of overdose in patients with opioid-inclusive substance use disorder diagnosis | 1/1/2010-12/31/2017
  Patient level regression controlling for year, age, sex, race, ethnicity
Predictors of opioid exposure (prescribing/dispending) and rate of neonatal abstinence syndrome for women of child-bearing age | 1/1/2010-12/31/2017
  Regression controlling for year, age, race, ethnicity at patient and 3-digit zip code level
Predictors of opioid-inclusive substance abuse disorder diagnosis and rate of neonatal abstinence syndrome for women of child-bearing age | 1/1/2010-12/31/2017
  Regression controlling for year, age, race, ethnicity at patient and 3-digit zip code level
Adjusted risk of emergency department and inpatient utilization in patients with opioid exposure (prescribing/dispensing) | 1/1/2010-12/31/2017
  Regression controlling for year, age, race, ethnicity at patient and 3-digit zip code level
Adjusted risk of emergency department and inpatient utilization in patients with opioid-inclusive substance abuse disorder diagnosis | 1/1/2010-12/31/2017
  Regression controlling for year, age, race, ethnicity at patient and 3-digit zip code level
Adjusted risk of emergency department and inpatient utilization in patients with opioid overdose diagnosis | 1/1/2010-12/31/2017
  Regression controlling for year, age, race, ethnicity at patient and 3-digit zip code level

SECONDARY OUTCOMES:
Characterization of opiate prescribing data for Guideline B patients | 1/1/2010-12/31/2017
  Count of patient encounters with opiate prescription record
Characterization of opiate dispensing data for Guideline B patients | 1/1/2010-12/31/2017
  Count of patient encounters with opiate dispensing record
Characterization of provider data for Guideline B patients | 1/1/2010-12/31/2017
  Count of providers from patient encounter records
Characterization of prescribing provider data for Guideline B patients | 1/1/2010-12/31/2017
  Count of providers from patient opiate prescribing records
Characterization of admitting source data for Guideline B patients | 1/1/2010-12/31/2017
  Count of patient encounters by admitting source type (frequencies)
Characterization of discharge disposition data for Guideline B patients | 1/1/2010-12/31/2017
  Count of patient encounters by discharge disposition type (frequencies)
Characterization of discharge status data for Guideline B patients | 1/1/2010-12/31/2017
  Count of patient encounters by discharge status (frequencies)
Characterization of facility data for Guideline B patients | 1/1/2010-12/31/2017
  Count of patient encounters by facility location/type (frequencies)
Characterization of urine drug screen data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patients with a urine drug screen lab result record
Characterization of urine drug screen results data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patients with a urine drug screen lab by result (frequencies)
Characterization of prescription type data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patient opiate prescriptions by RxNorm Term Types (frequencies)
Characterization of prescription dose data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patient opiate prescriptions by dose ordered unit of measure (frequencies)
Distribution of prescription dose data for Guideline B patients | 1/1/2010-12/31/2017
  Distribution of patient opiate prescriptions by dose ordered
Characterization of prescription dose frequency data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patient opiate prescriptions by dose frequency (frequencies)
Characterization of prescription supply data for Guideline B patients | 1/1/2010-12/31/2017
  Distribution of number of days supply of patient opiate prescriptions
Characterization of prescription quantity data for Guideline B patients | 1/1/2010-12/31/2017
  Distribution of prescription quantity for patient opiate prescriptions
Characterization of prescription refill data for Guideline B patients | 1/1/2010-12/31/2017
  Distribution of prescription refill numbers for patient opiate prescriptions
Characterization of procedure data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patient procedures by coding type (frequencies)
Characterization of vitals data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patient encounters with vitals records
Characterization of smoking/tobacco data for Guideline B patients | 1/1/2010-12/31/2017
  Counts of patient vital records by smoking/tobacco type (frequencies)
Characterization of language data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with language preference in record
Characterization of primary payer data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with primary payer data in record
Characterization of secondary payer data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with secondary payer data in record
Characterization of height data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with height data in record
Characterization of weight data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with weight data in record
Characterization of diastolic blood pressure data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with diastolic data in record
Characterization of systolic blood pressure data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with systolic data in record
Characterization of dispensed days supply data for Guideline B patients | 1/1/2010-12/31/2017
  Percent completeness of patients with days supply in the dispensing record

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A Lyman, JD, MHA, Principal Investigator — Louisiana Public Health Institute; Daniella Meeker, PhD, Principal Investigator — University of Southern California; Jason Doctor, PhD, Principal Investigator — University of Southern California
Locations (24):
- United States (24):
  - University of California - Irvine, Irvine, California
  - University of California - San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Los Angeles, Los Angeles, California
  - Patient-Centered SCAlable National Network for Effectiveness Research, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - San Mateo Medical Center, San Mateo, California
  - Health Choice Network, Miami, Florida
  - Research Action for Heath Network, New Orleans, Louisiana
  - University Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Health, Boston, Massachusetts
  - New York City Clinical Data Research Network, New York, New York
  - Weill Cornell Medicine, New York, New York
  - ADVANCE Clinical Data Research Network, Portland, Oregon
  - OCHIN, Inc, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - PaTH: Towards a Learning Health System Clinical Data Research Network, Pittsburgh, Pennsylvania
  - Veteran's Affairs Health System, Nashville, Tennessee
  - Baylor Scott & White Health, Dallas, Texas
  - University of Utah, Salt Lake City, Utah